CLINICAL TRIAL: NCT01383993
Title: An Open-Label, Non-Controlled, Multicenter, Intravenous To Oral Switch, Phase 2 Study To Evaluate The Pharmacokinetics, Safety And Tolerability Of Voriconazole In Immunocompromised Children Aged 2 To Less Than 15 Years Who Are At High Risk For Systemic Fungal Infection
Brief Title: Study Of The Pharmacokinetics And Safety Of Voriconazole In Children 2 To Less Than 15 Years Old Who Are At High Risk For Systemic Fungal Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A1501096
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Aspergillosis, Aspergilloma
Keywords: Open-Label; Pharmacokinetics; Intravenous to oral switch; Safety; Voriconazole; Immunocompromise; Children; High Risk For Systemic Fungal Infection
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 (Experimental): Immunocompromised children aged 2 to <15 and 12 to <15 years weighing <50 kg who are at high risk for systemic fungal infection.
  Interventions: Drug: Voriconazole
- 2.0 (Experimental): Immunocompromised children aged 12 to <15 years weighing more than 50 kg who are at high risk for systemic fungal infection.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Study Days 1: IV voriconazole 9 mg/kg q12h. Study Days 2 to 7: IV voriconazole 8 mg/kg q12h. Study Days 8 to 14: Oral voriconazole (POS) 9 mg/kg q12h with a maximum of 350 mg q12 h.
  Notes:
  If unable to switch to oral medication on Day 8, subjects can continue with IV treatment up to Day 20 before switching to oral dose.
  Only morning oral dose will be given on Day 14 (or the seventh day of oral dosing if IV regimen is extended). However, if clinically indicated, voriconazole treatment may be continued up to Day 30.
  (IV = Intravenous; POS = Powder for oral suspension)
  Other Names: UK-109,496; Vfend; Voriconazole
  Arms: 1.0
Drug: Voriconazole — Study Days 1: IV voriconazole 6 mg/kg q12h. Study Days 2 to 7: IV voriconazole 4 mg/kg q12h. Study Days 8 to 14: Oral voriconazole (POS) 200 mg q12h.
  Notes:
  If unable to switch to oral medication on Day 8, subjects can continue with IV treatment up to Day 20 before switching to oral dose.
  Only morning oral dose will be given on Day 14 (or the seventh day of oral dosing if IV regimen is extended). However, if clinically indicated, voriconazole treatment may be continued up to Day 30.
  (IV = Intravenous; POS = Powder for oral suspension)
  Other Names: UK-109,496; Vfend; Voriconazole
  Arms: 2.0

SUMMARY:
In this study we will measure the concentration of the drug called voriconazole which is used to fight infections caused by fungus in children who usually are cancer patients and have their immune system down. Since we know the dose in adults, and we think we know the matching doses in the young patients ages 2 to less than 15 years old, we will compare the amount of drug that goes into the system with what we know works in adults. We give the drug by a needle directly into the blood, then few days later we stop that and give the drug by mouth. Meanwhile, we draw a little bit of blood at certain times to measure the drug in it.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 2 to <15 years of age.
* Require treatment for the prevention of systemic fungal infection.
* Expected to develop neutropenia (ANC <500 cells/uL) lasting more than 10 days following chemotherapy.
* Anticipated to live for more than 3 months.

Exclusion Criteria:

* Evidence of any clinically significant liver or renal function or other abnormalities such as cardiac arrhythmia, hypokalemia, hypomagnesemia or hypocalcemia.
* Documented bacterial or viral infection not responding to appropriate treatment.
* Hypersensitivity to or severe intolerance of azole antifungal agents.
* Receiving other azoles or drugs that is are prohibited in the voriconazole label or associated.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Japan (6):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - National hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Sapporo Hokuyu Hosipital, Sapporo, Hokkaido
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi

REFERENCES:
- [Derived] Mori M, Kobayashi R, Kato K, Maeda N, Fukushima K, Goto H, Inoue M, Muto C, Okayama A, Watanabe K, Liu P. Pharmacokinetics and safety of voriconazole intravenous-to-oral switch regimens in immunocompromised Japanese pediatric patients. Antimicrob Agents Chemother. 2015 Feb;59(2):1004-13. doi: 10.1128/AAC.04093-14. Epub 2014 Dec 1. PMID 25451051
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501096&StudyName=Study%20Of%20The%20Pharmacokinetics%20And%20Safety%20Of%20Voriconazole%20In%20Children%202%20To%20Less%20Than%2015%20Years%20Old%20Who%20Are%20At%20High%20Risk%20For%20System

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Aged 2 to <12 Years: Immunocompromised children aged 2 to <12 years who are at high risk for systemic fungal infection. Voriconazole intravenous (IV) multiple dose (9 mg/kg on Day 1 and 8 mg/kg on Day 2 to 7 once every 12 hours) was administered in the morning and evening (up to Day 20 or more if clinically indicated). The oral dosing regimen (9 mg/kg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
- Participants Aged 12 to<15 Years and Weighed <50 kg: Immunocompromised children aged 12 to <15 years and weighed less than 50 kg who are at high risk for systemic fungal infection. Voriconazole intravenous (IV) multiple dose (9 mg/kg on Day 1 and 8 mg/kg on Day 2 to 7 once every 12 hours) was administered in the morning and evening (up to Day 20 or more if clinically indicated). The oral dosing regimen (9 mg/kg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
- Participants Aged 12 to<15 Years and Weighed ≥50 kg: Immunocompromised children aged 12 to <15 years and weighed greater than or equal to 50 kg who are at high risk for systemic fungal infection. Voriconazole intravenous (IV) multiple dose (6 mg/kg on Day 1 and 4 mg/kg on Day 2 to 7 once every 12 hours) was administered in the morning and evening (up to Day 20 or more if clinically indicated). The oral dosing regimen (200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Period: Overall Study
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Started | 15 | 4 | 2
Completed | 12 | 3 | 1
Not Completed | 3 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Marketed voriconazole in post-therapy | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg | Total
Number analyzed (Participants) | 15 | 4 | 2 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (2.8) | 12.5 (0.6) | 14.0 (0.0) | 9.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 1 | 12
  Male | 6 | 2 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Twelve Hours at Steady-State (AUC12,ss) Following IV Administration
Description: AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 7 (up to Day 20): predose, 1 hour after the start of infusion, 10-20 minutes after the end of infusion, and 4, 6, 8, and 12 hours after the start of infusion
Population: The pharmacokinetic parameter analysis was performed on all treated participants who had at least 1 of the pharmacokinetic parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
μg*h/mL | 51.92 (51) | 83.39 (56) | 17.27 (28)

2. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) Following IV Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
mcg/mL | 7.753 (38) | 9.233 (55) | 3.092 (42)

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following IV Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
hrs | 2.96 [0.950 to 4.00] | 4.00 [2.92 to 4.20] | 1.34 [1.00 to 1.67]

4. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Twelve Hours at Steady-State (AUC12,ss) Following Oral Administration
Description: AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
μg*h/mL | 48.23 (83) | 59.42 (67) | 10.00 (NA) — Number of analyzed participant was 1.

5. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) Following Oral Administration
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
mcg/mL | 7.755 (50) | 7.910 (45) | 2.030 (NA) — Number of analyzed participant was 1.

6. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) Following Oral Administration
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
hrs | 1.09 [0.917 to 3.78] | 1.00 [0.950 to 2.03] | 1.00 [1.00 to 1.00]

7. Primary Outcome: Number of Participants Assessed Near Distance Visual Acuity Test
Time Frame: Screening, Day 7 (the 7th day of IV treatment), Day 8 (the 1st day of oral treatment), Day 14 (the 7th day of oral treatment), and the 30-day follow-up visit
Population: The safety analysis was performed on all subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- All Participants: Immunocompromised children aged 2 to <15 years who are at high risk for systemic fungal infection. Voriconazole intravenous (IV) multiple dose (9 mg/kg or 6 mg/kg on Day 1 and 8 mg/kg or 4 mg/kg on Day 2 to 7 once every 12 hours) was administered in the morning and evening (up to Day 20 or more if clinically indicated). The oral dosing regimen (9 mg/kg or 200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | All Participants
Number analyzed (Participants) | 21
participants
  Screening | 18
  The 7th day of IV treatment | 18
  The 1st day of oral treatment | 17
  The 7th day of oral treatment | 15
  The 30 day follow up visit | 14

8. Primary Outcome: Number of Participants Assessed Color Vision Test
Time Frame: as for outcome 7
Population: The safety analysis was performed on all subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 21
participants
  Screening | 19
  The 7th day of IV treatment | 18
  The 1st day of oral treatment | 17
  The 7th day of oral treatment | 15
  The 30 day follow up visit | 14

9. Primary Outcome: Number of Participants Assessed Visual Questionnaire
Time Frame: as for outcome 7
Population: The safety analysis was performed on all subjects who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 21
participants
  Screening | 19
  The 7th day of IV treatment | 18
  The 1st day of oral treatment | 17
  The 7th day of oral treatment | 15
  The 30 day follow up visit | 14

10. Secondary Outcome: Ratio of AUC12,ss Following IV Administration Relative to AUC12,ss Following Oral Administration
Description: Ratio was calculated from the following formula; AUC12,ss Following Oral Administration over AUC12,ss Following IV Administration
Time Frame: AUC12, ss for IV:Day 7 (up to Day 20): predose, 1 hour after the start of infusion, 10-20 minutes after the end of infusion. AUC12,ss for oral: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
ratio | 1.077 (0.547) | 0.648 (0.015) | 0.476 (NA) — Number of analyzed participant was 1.

11. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Twelve Hours at Steady-State (AUC12,ss) of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Description: AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
μg*h/mL | 66.50 (30) | 80.99 (41) | 40.00 (2)

12. Secondary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
mcg/mL | 6.381 (28) | 8.066 (34) | 3.835 (1)

13. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 4 | 2
hrs | 5.05 [2.87 to 11.8] | 4.49 [1.00 to 11.1] | 3.84 [1.67 to 6.00]

14. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Twelve Hours at Steady-State (AUC12,ss) of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Description: AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
μg*h/mL | 79.86 (36) | 90.84 (19) | 34.40 (NA) — Number of analyzed participant was 1.

15. Secondary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
mcg/mL | 7.971 (31) | 8.912 (22) | 3.720 (NA) — Number of analyzed participant was 1.

16. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 14 (the 7th day of oral treatment) or later: predose, and 1, 2, 4, 6, 8, and 12 hours after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Number analyzed (Participants) | 14 | 3 | 1
hrs | 2.07 [0.000 to 7.78] | 2.03 [0.950 to 4.00] | 3.80 [3.80 to 3.80]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Participants Aged 2 to <12 Years | Participants Aged 12 to<15 Years and Weighed <50 kg | Participants Aged 12 to<15 Years and Weighed ≥50 kg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 13/15 | 4/4 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Aged 2 to <12 Years (N=15) | Participants Aged 12 to<15 Years and Weighed <50 kg (N=4) | Participants Aged 12 to<15 Years and Weighed ≥50 kg (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 2 | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0 | 0
Colour blindness (Congenital, familial and genetic disorders) | 1 | 0 | 0
Chromatopsia (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 5 | 3 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Hyperaemia (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.